CLINICAL TRIAL: NCT04734808
Title: EEG Brain Activity During A Progressive Cycling Protocol
Brief Title: EEG Brain Activity At Various Cycling Intensities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University Maribor (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Marusic, Dr. Uroš Marušič, Science and Research Centre Koper
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: TwinBrainCycling
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: EEG; Brain Imaging; Brain Waves; Cycling; Intensity
MeSH Terms: interventions — Electroencephalography; Electromyography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electroencephalography — Electroencephalography is an electrophysiological monitoring method to record electrical activity of the brain.
  Other Names: EEG
Diagnostic Test: Electromyography — Electromyography is an electrodiagnostic medicine technique for evaluating and recording the electrical activity produced by skeletal muscles. We will use the hdEMG version.
  Other Names: hdEMG

SUMMARY:
The aim of this study is to investigate brain activity with EEG during incremental cycling at various cycling intensities.

DETAILED DESCRIPTION:
Increases in EEG power spectra have been found during graded cycling to fatigue linking brain activity to exercise intensity. Additionally, to the activation of the classical motor control regions (e.g.: motor, somatosensory, premotor and supplementary motor cortices and cerebellum), the activation of the regions associated with autonomic regulation (i.e.: insular cortex) during exercise, as well as reduced activation of cognitive-related areas (i.e.: prefrontal cortex), an effect that increased at higher perceived intensities of cycling has been observed.

Furthermore, the precentral gyrus and cerebellar vermis, as well as brain areas (e.g.: posterior cingulate cortex (PCC) and precuneus) have been associated with higher levels of perceived exertion as well. Although the results were assessed sing a specially designed compatible fMRI cycling ergometer (Fontes et al., 2020), due to which the brain imaging techniques were limited to static (and horizontal) measurement conditions during cycling, we believe that the present study clearly distinguishes between claims proposed by different theoretical frameworks on brain responses during exercise.

Therefore, the aim of this study is to examine the brain activity with EEG during the same incremental protocol, which will allow us to investigate the functioning of surface electrocortical activation patterns during progressive cycling exercise. Furthermore, using the advanced brain image analysis (machine learning techniques and standardized low-resolution electromagnetic tomography - sLORETA) helped us determine the frequency spectrum of brain activity in the same brain areas.

ELIGIBILITY:
Inclusion Criteria:

* Heathy and recreationaly active men
* No significant muscular, skeleton or nervous system damage
* Cycloergometry test (positive)

Exclusion Criteria:

* Nervous system disorders
* Cardiovascular disorders (e.g.: high blood pressure, arrhythmia...)
* Asthma

Ages: 22 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Beta band suppression | During the intervention
  Reduction of beta is one of the cortical markers which is usually obtained from the central electrodes and occurs with movement initiation.

SECONDARY OUTCOMES:
Brain mapping | During the intervention
  Analyzing the change in (de)activated "regions of interest" (ROI) of the brain between cycling during increasing exercise conditions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maribor, Maribor, Slovenia

REFERENCES:
- [Background] Bailey SP, Hall EE, Folger SE, Miller PC. Changes in EEG during graded exercise on a recumbent cycle ergometer. J Sports Sci Med. 2008 Dec 1;7(4):505-11. eCollection 2008. PMID 24149958
- [Background] Fontes EB, Bortolotti H, Grandjean da Costa K, Machado de Campos B, Castanho GK, Hohl R, Noakes T, Min LL. Modulation of cortical and subcortical brain areas at low and high exercise intensities. Br J Sports Med. 2020 Jan;54(2):110-115. doi: 10.1136/bjsports-2018-100295. Epub 2019 Aug 16. PMID 31420319
- [Background] Fontes EB, Okano AH, De Guio F, Schabort EJ, Min LL, Basset FA, Stein DJ, Noakes TD. Brain activity and perceived exertion during cycling exercise: an fMRI study. Br J Sports Med. 2015 Apr;49(8):556-60. doi: 10.1136/bjsports-2012-091924. Epub 2013 Jun 1. PMID 23729175
- [Background] Enders H, Cortese F, Maurer C, Baltich J, Protzner AB, Nigg BM. Changes in cortical activity measured with EEG during a high-intensity cycling exercise. J Neurophysiol. 2016 Jan 1;115(1):379-88. doi: 10.1152/jn.00497.2015. Epub 2015 Nov 4. PMID 26538604